CLINICAL TRIAL: NCT02176759
Title: Iron Absorption From Rice Fortified With Ferric Pyrophosphate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Rice_SFePP
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-06

CONDITIONS: Iron Deficiency; Anemia; Iron Deficiency Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia; Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Regular FePP (Experimental): Rice (50g dry weight) fortified with 4mg regular FePP
  Interventions: Other: Administration of rice fortified with regular FePP
- Regular FePP with citrate added during extrusion (Experimental): Rice (50g dry weight) fortified with 4mg regular FePP and citrate added during the extrusion process
  Interventions: Other: Administration of rice fortified with regular FePP with citrate added during extrusion
- Regular FePP with citrated added at consumption (Experimental): Rice (50g dry weight) fortified with 4mg regular FePP and citrate shortly added before consumption
  Interventions: Other: Administration of rice fortified with regular FePP and citrate added at consumption
- Ferrous sulphate (Active Comparator): Rice (50g dry weight) fortified with 4mg ferrous sulphate
  Interventions: Other: Administration of rice fortified with ferrous sulphate

INTERVENTIONS:
Other: Administration of rice fortified with regular FePP
  Arms: Regular FePP
Other: Administration of rice fortified with regular FePP with citrate added during extrusion
  Arms: Regular FePP with citrate added during extrusion
Other: Administration of rice fortified with regular FePP and citrate added at consumption
  Arms: Regular FePP with citrated added at consumption
Other: Administration of rice fortified with ferrous sulphate
  Arms: Ferrous sulphate

SUMMARY:
Ferric pyrophosphate (FePP) is a water-insoluble, food grade iron compound used to fortify rice, infant cereals and chocolate-drink powders as it causes no organoleptic changes to the food vehicle. However, it is only of low absorption in man. Therefore, strategies to enhance the bioavailability of FePP, such as adding citrate or decreasing the particle size of FePP need to be investigated. The primary objectives of the present study are: 1) to test whether the presence of citrate in iron fortified rice with FePP results in higher iron bioavailability, and 2) to test whether the presence of citrate in the rice grain during the extrusion and cooking process results in higher iron bioavailability compared with iron-fortified rice where citrate has been added shortly before consumption. As a secondary objective the investigators will compare the absorption from different FePP combinations with a reference meal fortified with ferrous sulphate. The investigator hypothesize that the addition of citrate enhances iron absorption and that the positive effect is greater when the citrate is added during the extrusion.

The investigator will conduct an iron absorption study in 20 women, 18 to 45 years old to evaluate the iron bioavailability from extruded rice fortified with 1) regular FePP, 2) regular FePP and citrate (both extruded into the rice kernels), 3) regular FePP and citrate added at the time of consumption, and 4) from normal rice fortified with ferrous sulphate at the time of consumption. Iron absorption will be measured as erythrocyte incorporation of stable iron isotopes at least 14 days after the administration of the isotopically labelled test meals. The iron absorption from the different meals within the same participant will be compared by repeated-measures ANOVA followed by a Bonferroni corrected pairwise comparison.

The present study will provide important data where iron bioavailability from rice is accurately and directly measured using stable isotopic labels as absorption tracers. This direct data can be used to base decisions on the level of fortification, can potentially reduce costs and optimize iron delivery to the targeted population in iron fortification programs.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* Normal body Mass Index (18.5 - 25 kg/m2)
* Body weight < 65 kg
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by a pregnancy test)
* Lactating
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using Fe stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 2 | baseline, 2 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 2 in the isotopic ratio of iron in blood at week 4 | 2 weeks, 4 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.
Change from week 4 in the isotopic ratio of iron in blood at week 6 | 4 weeks, 6 weeks
  The change in the isotopic ratio of iron will be measured after the administration of test meal including iron isotopes.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Hackl L, Speich C, Zeder C, Sanchez-Ferrer A, Adelmann H, de Pee S, Tay F, Zimmermann MB, Moretti D. Cold Extrusion but Not Coating Affects Iron Bioavailability from Fortified Rice in Young Women and Is Associated with Modifications in Starch Microstructure and Mineral Retention during Cooking. J Nutr. 2017 Dec;147(12):2319-2325. doi: 10.3945/jn.117.259085. Epub 2017 Oct 18. PMID 29046406
- [Derived] Hackl L, Cercamondi CI, Zeder C, Wild D, Adelmann H, Zimmermann MB, Moretti D. Cofortification of ferric pyrophosphate and citric acid/trisodium citrate into extruded rice grains doubles iron bioavailability through in situ generation of soluble ferric pyrophosphate citrate complexes. Am J Clin Nutr. 2016 May;103(5):1252-9. doi: 10.3945/ajcn.115.128173. Epub 2016 Apr 6. PMID 27053382